CLINICAL TRIAL: NCT04928755
Title: Design and Evaluation of a Novel Methodology for Stereotactic Ablative Radiotherapy for Lung Cancer: Reducing Treatment Side-effects and Enabling More Patients to Benefit From This Treatment
Brief Title: Design and Evaluation of a Novel Methodology for SABR for Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19ONCN262953
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
Keywords: Radiotherapy; SABR
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aims: To increase the number of patients that benefit from Stereotactic Ablative Radiotherapy (SABR) for lung cancer using new treatment methods that reduce the amount of non-cancer tissue receiving a high radiation dose without affecting tumour dose coverage.

Background: SABR is a treatment for lung cancer which offers major advantages over conventional radiotherapy. It is a more precise highly effective treatment with significantly improved treatment outcomes (greater elimination of cancer cells).

SABR requires high doses per treatment so extreme accuracy is required to minimise healthy tissue damage. Normal breathing results in significant tumour movement, therefore to avoid missing the tumour, larger volumes need to be treated, resulting in more good tissue damage.

UK Standard practice requires the tumour to be irradiated in all positions during breathing whilst the new approach targets the tumours at the position it spends most time to minimise normal tissue affected by radiation.

Current practice for SABR patients would be improved (fewer severe radiation side-effects) and potentially could become a viable treatment for high risk patients.

Methods: 30 SABR patients receiving current standard SABR treatment will be recruited. This is an observation study in which patients will continue to receive standard of care but in addition:

* A camera will be used to make videos of how the patient's chest moves in 3D at CT and treatment. I will build a complex mathematical model that infers movement of the tumour from movement of the chest.
* Their breathing patterns, corresponding tumour motions and treatments plans will be utilised to develop a method for safely implementing the new treatment approach.

ELIGIBILITY:
Inclusion Criteria:

All patients eligible for and who have consented to receive Lung SABR at the Royal Surrey County Hospital will be eligible for entry into this study.

• Over 18 years old (radiotherapy is not delivered to 16-18yr olds at RSFT). No upper age limit.

Exclusion Criteria:

Patients with irregular breathing motion resulting in failed 4DCT

* Patients with unusual chest surface deformities
* Patients who lack the capacity to consent
* Patients unable to read and communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving SABR Lung Radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Design a methodology that ensures tumour dose coverage is obtained when using the new treatment approach. | 2 years

SECONDARY OUTCOMES:
Use a novel markerless non-contact approach (Microsoft Kinect) to create a model to correlate external respiratory motion with internal tumour motion. | 2years
Validate and refine correlation between predicted tumour motion and actual breathing motion. | 2years

IPD SHARING:
Plan to Share IPD: No